CLINICAL TRIAL: NCT06579508
Title: Effects of High-intensity Intermittent Exercise With Recovery Hypoxia and Taurine Supplementation in Women With Obesity on Metabolic and Mitochondrial Parameters
Brief Title: Effects of High-intensity Exercise With Hypoxia and Taurine Supplementation on Metabolic and Mitochondrial Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hypoxia_Taurine
Record Dates: First submitted 2024-08-20; First posted 2024-08-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: Mitochondrial disfunction; Oxidative stress; Inter-effort Hypoxia; Physical Exercise; Obesity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Off-Road Motor Vehicles

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Masking Description: Participants will be randomly distributed into 5 groups:
  Control; Normoxia + placebo (Nor-P); Normoxia + taurine (Nor-T); Hypoxia + placebo (Hyp-P); Hypoxia + Taurine (Hyp-T). Control group is the only group without training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): No intervention, only the evaluations will be done.
- Normoxia - Placebo (Placebo Comparator): High-intensity interval cycle ergometer train, with inter effort normoxia (FiO2 = 21%).
  Interventions: Other: Cycle ergometer
- Normoxia - Taurina (Placebo Comparator): High-intensity interval cycle ergometer train, with inter effort normoxia (FiO2 = 21%).
  Interventions: Other: Cycle ergometer
- Hypoxia - Placebo (Placebo Comparator): High-intensity interval cycle ergometer train, with inter effort hypoxia (FiO2 = 12%).
  Interventions: Other: Cycle ergometer
- Hypoxia - Taurina (Experimental): High-intensity interval cycle ergometer train, with inter effort hypoxia (FiO2 = 12%).
  Interventions: Other: Cycle ergometer

INTERVENTIONS:
Other: Cycle ergometer — The initial part will last 5 minutes at low intensity, corresponding to "easy" by the RPE.
  The main part will be performed at the intensity of training zone 3 (100-110% of the Lan), lasting 5 minutes with a rest of 2.5 minutes between exercises. The intensity will be controlled by HR and RPE.
  The final part will last 3 minutes at low intensity, corresponding to "easy" by the RPE.
  The load progression occurred during the first four weeks, starting with 3 sets and adding 1 set per week.
  The intensity of each effort is 100-110%HRAnTh.
  Other Names: Bike
  Arms: Hypoxia - Placebo; Hypoxia - Taurina; Normoxia - Placebo; Normoxia - Taurina

SUMMARY:
The prevalence of obesity in Brazil is one of the highest in Latin America. As an inflammatory disease, obesity needs to be treated, and one of the best interventions is exercise. This research aims to learn more about the effects of combining high-intensity training, recovery hypoxia, and taurine supplementation. To better understand these effects, the researchers will compare hypoxia and normoxia, as well as taurine and placebo, with all participants training in the same way. The researchers will also investigate mitochondrial respiration and food consumption to connect certain aspects of obesity with overall health.

DETAILED DESCRIPTION:
Obesity is characterized by a chronic inflammatory state, often linked with elevated oxidative stress and mitochondrial dysfunction. While physical exercise can trigger inflammatory responses due to muscle damage, it also promotes significant bodily adaptations, particularly in body composition, physical fitness, and skeletal muscle tissue, including enhanced mitochondrial dynamics. Moderate hypoxia, when combined with exercise, further amplifies these benefits by increasing the expression of genes related to mitochondrial biogenesis, GLUT1 expression, and angiogenesis. Previous findings suggest that high-intensity physical activity not only improves cardiorespiratory capacity and alters body composition but also significantly elevates inflammation. Consequently, taurine, a supplement known for its anti-inflammatory properties and ability to reduce oxidative stress, should be considered to mitigate these issues and optimize the benefits of exercise and hypoxia. Based on these premises, it is hypothesized that the combination of taurine supplementation with physical training under recovery hypoxia may reduce the significant rise in pro-inflammatory cytokines, thereby enhancing the potential benefits of exercise and moderate hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age between 25 - 45 years old;
* BMI between 30 - 35kg/m²;
* Not be on a diet;
* Not be on a physical activity program;
* Not be menopaused.

Exclusion Criteria:

* Smokers;
* Alcoholics;
* Use thyroid medication;
* Carry out nutritional monitoring or in treatment for weight loss;
* Hypertension;
* Metabolical syndrome;
* Have any comorbidity associated to obesity;
* Drugs use.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Anthropometry - Height | 12 weeks
  Dual energy x-ray absorptiometry (DEXA) will be use for:
  Height measured in meters.
Anthropometry - Weight | 12 weeks
  Dual energy x-ray absorptiometry (DEXA) will be use for:
  Changes in body weight in kilograms (kg).
Anthropometry - BMI | 12 weeks
  Dual energy x-ray absorptiometry (DEXA) will be use for:
  Changes in body mass index (BMI = weight measured(kg) / (height (m)²).
Body composition - Free-fat mass | 12 weeks
  Dual energy x-ray absorptiometry (DEXA) will be use for:
  Changes in body composition for fat-free mass (grams and %).
Body composition - Fat mass | 12 weeks
  Dual energy x-ray absorptiometry (DEXA) will be use for:
  Changes in body composition for fat mass (grams and %).
Body composition - Bone | 12 weeks
  Dual energy x-ray absorptiometry (DEXA) will be use for:
  Changes in body composition for bone mineral content (g.cm²).
Lipid profile - Cholesterol | 12 weeks
  Quantified by Total Liquiform Cholesterol Kit, HDL Cholesterol Kit and Liquiform Triglycerides Kit, from Labtest diagnóstica®, using an enzymatic system and absorbance spectrophotometer:
  Changes in total cholesterol (mg/dL).
Lipid profile - Triglycerides | 12 weeks
  Quantified by Total Liquiform Cholesterol Kit, HDL Cholesterol Kit and Liquiform Triglycerides Kit, from Labtest diagnóstica®, using an enzymatic system and absorbance spectrophotometer:
  Changes in triglycerides (mg/dL).
Lipid profile - HDL/LDL | 12 weeks
  Quantified by Total Liquiform Cholesterol Kit, HDL Cholesterol Kit and Liquiform Triglycerides Kit, from Labtest diagnóstica®, using an enzymatic system and absorbance spectrophotometer:
  Changes in HDL-cholesterol and LDL-cholesterol (mg/dL).
Lipid profile - Glucose | 12 weeks
  Quantified by Total Liquiform Cholesterol Kit, HDL Cholesterol Kit and Liquiform Triglycerides Kit, from Labtest diagnóstica®, using an enzymatic system and absorbance spectrophotometer:
  Changes in blood glucose (mg/dL).
Inflammatory profile - pro inflammatory | 12 weeks
  Changes in serum levels of cytokines will be evaluated with MILLIPLEX® Kit. Pro- inflammatory citokines: IL-6, TNF-α (pg/mL).
Inflammatory profile - anti inflammatory | 12 weeks
  Changes in serum levels of cytokines will be evaluated with MILLIPLEX® Kit. Ant- inflammatory citokines: IL-10 (pg/mL), Adiponectin (ng/mL).
Aerobic performance - HRAnTh | 12 weeks
  Physical tests performed pre-, after 6 weeks and post- intervention to assess aerobic physical fitness by incremental test in cycle ergometer. The test aim to evaluate:
  Anaerobic threshold (AT) using heart rate (HR).
Aerobic performance - IAnTh | 12 weeks
  Physical tests performed pre-, after 6 weeks and post- intervention to assess aerobic physical fitness by incremental test in cycle ergometer. The test aim to evaluate:
  Anaerobic threshold (AT) using intensity in Watts (W).
Aerobic performance - RPEAnTh | 12 weeks
  Physical tests performed pre-, after 6 weeks and post- intervention to assess aerobic physical fitness by incremental test in cycle ergometer. The test aim to evaluate:
  Anaerobic threshold (AT) using Rate of Perceived Effort (RPE).
Aerobic performance - LacAnTh | 12 weeks
  Physical tests performed pre-, after 6 weeks and post- intervention to assess aerobic physical fitness by incremental test in cycle ergometer. The test aim to evaluate:
  Anaerobic threshold (AT) using lactate concentration [lac-].
Aerobic performance - VO2 | 12 weeks
  Physical tests performed pre-, after 6 weeks and post- intervention to assess aerobic physical fitness by incremental test in cycle ergometer. The test aim to evaluate:
  VO2peak in ml.kg-1.min-1.
Food Intake | 12 weeks
  A food record of three non-consecutive days: two days of the week and one day in the weekend. This evaluation will last 12 weeks. Will be evaluated with Dietwin® software (São Paulo, Brazil):
  The macronutrients, micronutrients and fiber in quilocalories and percentage (%)
Food quality | 12 weeks
  The feed will undergo analysis through the NOVA Classification. By NOVA, food will be classified into four groups: Group 1 - Unprocessed or minimally processed foods; Group 2 - Processed culinary ingredients; Group 3 - Processed foods; Group 4 - Ultra-processed foods.
  For each category, the total calories ingested will be calculated, and later, represented in percentage (%) the participation of each food group in the general diet.
Taurine rates | 12 weeks
  The participants will supplement 3g of taurina or placebo during 12 weeks. The rate of plasmatic taurine (mmol) will be evaluated during pre and post intervention.
Muscle biopsy - RNA | 12 weeks
  After biopsy the tissue will be treated for:
  qPCR analysis.
Muscle biopsy - Protein | 12 weeks
  After biopsy the tissue will be treated for:
  Western blotting analysis.
Muscle biopsy - Mitochondria | 12 weeks
  After biopsy the tissue will be treated for:
  High-resolution respirometry of muscle fibers analysis.

SECONDARY OUTCOMES:
Training measures - RPE | 12 weeks
  The Borg scale will be use to quantify the:
  Rate of Perceived Effort (RPE) - will be noted after each effort during all the training program.
Training measures - TRIMP | 12 weeks
  The internal load will be calculated using TRIMP:
  Calculated multipling the RPE for the time in effort (TRIMP = RPE * time in effort), for each participant and training session.
Training measures - SP02 | 12 weeks
  The Oxygen saturation (SpO2) will be measure in percent (%), using a pulse oximeter.
  SpO2 (%) will be noted after the end of the effort, the lowest point during the rest and in the end of the rest.
Training measures - HR | 12 weeks
  The heart rate (HR) will be measure in beats per minute (BPM) with Polar clock.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela C Viliod, Principal Investigator — USP
Locations (2):
- Brazil (2):
  - University of São Paulo, School of Physical Education and Sports of Ribeirão Preto., Ribeirão Preto, São Paulo
  - University of São Paulo, School of Physical Education and Sports of Ribeirão Preto, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No